CLINICAL TRIAL: NCT00459732
Title: Zinc and Bone Metabolism in Thalassemia
Brief Title: Zinc & Bone Health in Thalassemia: The Think Zinc Study
Acronym: ThinkZn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Children's Hospital of Philadelphia (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004-106; K23HL076468 (NIH); NCT00480415 (obsolete NCT alias)
Record Dates: First submitted 2007-04-11; First posted 2007-04-12 (Estimated); Results first posted 2011-09-30 (Estimated); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Thalassemia
Keywords: zinc, thalassemia, bone mineral density
MeSH Terms: conditions — Thalassemia | interventions — Zinc; Zinc Sulfate; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Capsule (Placebo Comparator): placebo capsule, similar in size, shape and color to zinc capsule, taken once daily for 18 months
  Interventions: Dietary Supplement: Placebo
- Zinc (25 mg/d) (Active Comparator): 25 mg of elemental Zinc as zinc sulphate taken once daily for 18 months
  Interventions: Dietary Supplement: Zinc

INTERVENTIONS:
Dietary Supplement: Zinc — 25 mg of elemental zinc as zinc sulphate take once daily for 18 months
  Other Names: zinc sulphate; elemental zinc
  Arms: Zinc (25 mg/d)
Dietary Supplement: Placebo — Placebo capsule, identical to the zn capsule in size, shape and color, taken once daily for 18 months
  Other Names: "sugar" pill
  Arms: Placebo Capsule

SUMMARY:
The purpose of this study is to test whether zinc can improve bone health in young patients with thalassemia.

DETAILED DESCRIPTION:
The primary aim of this study is to determine if zinc supplementation improves bone health in young patients with thalassemia. Osteoporosis is a significant co-morbidity in patients with thalassemia which leads to decreased quality of life. The most effective way to prevent osteoporosis is to build strong, dense bones in the early years. A combination of disease, endocrine and nutritional factors likely contribute to the etiology of osteoporosis in this population. However, even well transfused patients with normal gonadal function who are supplemented with calcium have low bone mass. It is hypothesized that patients with thalassemia have low bone mass, in part, due to zinc deficiency. Sub-optimal zinc status has been identified in patients with thalassemia and zinc supplementation has been shown to improve linear growth. To test the primary hypothesis, an 18 month randomized placebo-controlled trial of zinc supplementation (25 mg Zn/day) vs. placebo will be conducted in 60 young patients (6-30 yrs) with thalassemia and low bone mass (spine BMD Z-score <-1.0). Bone health, as estimated from measurements of bone mass (by DXA and pQCT) and markers of bone formation and resorption will be the primary outcome variables. This will be the first study to examine the effects of zinc. supplementation on bone health in patients with thalassemia. If zinc supplementation is found to have a clinically important effect, this simple, safe, non-invasive therapy could quickly become a part of the standard care of these young patients and improve overall health in children and adult patients with thalassemia

ELIGIBILITY:
Inclusion Criteria:

* 6 to 30 years of age
* thalassemia
* bone mineral density Z-score < -1.0 (by DXA)

Exclusion Criteria:

* Bone marrow transplant recipient
* Currently prescribed treatment for low bone mass other than calcium or vitamin D (e.g. calcitonin, bisphosphonates)
* Currently prescribed zinc supplementation who are unable or unwilling to stop during this trial
* Currently participating in another trial with a medication known to affect bone mineral density.
* Chronic use of systemic corticosteroids
* Untreated hypogonadism or growth hormone deficiency
* Baseline serum copper < 70 µg/dL
* Baseline vitamin D-25OH < 11 ng/mL
* Pregnant or lactating at study entry

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2006-04; Primary Completion 2009-10 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen B. Fung, PhD, RD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (3):
- United States (3):
  - Children's Hospital & Research Center, Oakland, Oakland, California
  - University of California, San Francisco, San Francisco, California
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Fung EB, Kwiatkowski JL, Huang JN, Gildengorin G, King JC, Vichinsky EP. Zinc supplementation improves bone density in patients with thalassemia: a double-blind, randomized, placebo-controlled trial. Am J Clin Nutr. 2013 Oct;98(4):960-71. doi: 10.3945/ajcn.112.049221. Epub 2013 Aug 14. PMID 23945720

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 3 hematology clinics in the US between April, 2006 and May, 2008. 114 potentially eligible patients were screened, 43 were considered eligible and consented to participation.
Pre-assignment Details: Following enrollment, prior to group assignment, subjects were screened for copper and vitamin D status. If serum copper was <70ug/dL and/or 25OH vitamin D <20ng/mL, they were placed on daily supplementation, 2 mg Cu/day and/or 1000 IU vitamin D/day.
Groups:
- Zinc: 25 mg of zinc as zn sulfate taken daily
- Placebo: daily capsule similar in size/color to zn was taken daily by this group
Period: Overall Study
Arm/Group | Zinc | Placebo
Started | 23 | 17
Completed | 19 (4 on zn dropped: 1 pregnant and 1 nausea after baseline, 1 lost to followup, 1 exited after 12 month) | 14 (3 on placebo dropped: 1 pregnant after 12 mo, 1 lost to followup, one died after 12 month timepoint)
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zinc | Placebo | Total
Number analyzed (Participants) | 23 | 17 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 9 | 19
  Between 18 and 65 years | 13 | 8 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.7 (5.6) | 17.4 (4.9) | 17.6 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 11 | 8 | 19
Region of Enrollment [Number; unit: participants]
  United States | 23 | 17 | 40
Plasma Zinc [Mean (Standard Deviation); unit: mcg/dL] — Concentration of zinc within the plasma at baseline, mcg/dL
  mcg/dL | 77 (11) | 79 (14) | 78 (12)
Spine Z-score [Mean (Standard Deviation); unit: Z-score] — Spine standard deviation score (Z-score) determined by baseline DXA bone density scan
  Z-score | -1.9 (1.0) | -2.4 (1.1) | -2.1 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Lumbar Spine Bone Mineral Density (BMD) by DXA (Baseline to 18 Months)
Description: Change in pa spine bone mineral density by DXA between baseline and 18 months
Time Frame: 0 to 18 months
Population: Intention to treat analysis of all subjects who completed the protocol in each arm of the study (zinc vs. placebo).
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Zinc | Placebo
Number analyzed (Participants) | 18 | 14
Percent Change | 5.9 (5.3) | 1.5 (9.0)
Statistical Analysis 1: Comparison: Zinc vs Placebo; Test type: Superiority or Other; p = 0.13, ANOVA

2. Primary Outcome: Change in Whole Body Bone Mineral Content (BMC) by DXA (Baseline to 18 Months)
Time Frame: Baseline to 18 months
Population: Intention to treat analysis in those who completed the 18 month timepoint (zinc vs. placebo)
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Zinc | Placebo
Number analyzed (Participants) | 17 | 14
Percent change | 6.1 (6.1) | 2.2 (9.2)
Statistical Analysis 1: Comparison: Zinc vs Placebo; Test type: Superiority or Other; p = 0.44, ANOVA; Repeated measures

3. Secondary Outcome: Osteocalcin, a Marker of Bone Formation
Description: Absolute change in serum osteocalcin between 0 and 18 months, intention to treat analysis between the zinc and placebo groups
Time Frame: Baseline to 18 months
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Zinc | Placebo
Number analyzed (Participants) | 19 | 14
ng/mL | 8.8 (17.1) | -4.3 (23.2)
Statistical Analysis 1: Comparison: Zinc vs Placebo; Test type: Superiority or Other; p = 0.16, ANCOVA; Repeated measures analysis of variance adjusted for baseline osteocalcin level

ADVERSE EVENTS:
Time Frame: Recorded between baseline and 18 month time point (end of study)
Description: Adverse events were collected at 5 timepoints, 3, 6, 12 and 18 months after start of supplementation.
Arm/Group | Zinc | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/17
Other Adverse Events (participants affected / at risk) | 17/19 | 8/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zinc (N=23) | Placebo (N=17)
Death (Cardiac disorders) | 0 (0) | 1 (1) — One subject on the placebo arm of the trial died from cardiomyopathy secondary to iron overload after the 12 month time point.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zinc (N=19) | Placebo (N=14)
Nausea (Gastrointestinal disorders) | 10 (14) | 8 (10)
Diarrhea (Gastrointestinal disorders) | 3 (7) | 5 (7)
Stomach Upset (Gastrointestinal disorders) | 11 (13) | 8 (11) — Includes general stomach upset and/or cramping
Fatigue (Blood and lymphatic system disorders) | 5 (6) | 5 (6) — Fatigue that is different that usual pre-transfusion fatigue
Headache (Nervous system disorders) | 8 (9) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No